CLINICAL TRIAL: NCT01070849
Title: Effect and Sustainability of a Bio-psycho-social Exercise Program (RÜCKGEWINN) for Chronic Low Back Pain in Rehabilitation Aftercare - a Randomised Controlled Trial
Brief Title: A Bio-psycho-social Exercise Program (RÜCKGEWINN) for Chronic Low Back Pain in Rehabilitation Aftercare
Acronym: RÜCKGEWINN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: Deutsche Rentenversicherung (Other)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Chair for Exercise and Health, University of Erlangen-Nürnberg
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 8011 - 106 - 31/31.87
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Low Back Pain
Keywords: exercise; physical activity
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- a) educational booklet (Active Comparator)
  Interventions: Other: educational booklet
- b) IRENA (Active Comparator)
  Interventions: Other: IRENA
- c) RÜCKGEWINN (Experimental)
  Interventions: Other: RÜCKGEWINN

INTERVENTIONS:
Other: educational booklet — Participants will receive an educational booklet and the advice to return to normal activities as soon as possible from their rehabilitation practitioner in their dismissal examination. As educational booklet the German version of the "back book" of Burton et al. was chosen. This booklet provides information about the new approach to back pain, causes of back pain, dealing with an attack of back pain, risk factors for development of chronic back pain and the role of activity. All information that is provided is in accordance with actual scientific knowledge and is based on a bio-psycho-social model of back pain like described in Waddell.
  Arms: a) educational booklet
Other: IRENA — Participants will be introduced into the normal IRENA program (in German: Intensivierte Rehabilitationsnachsorge), which is usual care in Germany. Every patient will be assigned to a certified aftercare facility near their residential area. Aftercare practitioners and patients can compile an individual therapeutic package from certain appointed therapeutic services. Predominantly resistance training, gymnastics, aquatic exercise, back school and recreation exercises are prescribed by the physicians for aftercare. Most therapies are carried out in open access groups of at least 6 patients without being specific for medical indication. In the IRENA program it is possible to pass the intended 24 exercise sessions with different frequency per week. Usually participants do two or three exercise sessions per week with duration of 90 to 120 minutes per session. Every aftercare facility offers certain therapy combinations at different days in week.
  Arms: b) IRENA
Other: RÜCKGEWINN — For long term sustainability and the enhancement of intensity of the rehabilitation process this investigational aftercare intervention shows formal and didactic divergences from standard programmes in rehabilitation aftercare. Three important areas for multidimensional interventions are targeted: attitude and behaviour change concerning back pain, guidance to health enhancing physical activity, improvement of health related physical fitness. Every 90 minutes taking exercise session contains parts for mediation of knowledge, for behavioural modulation and for physical exercises and interlocks them in the mediation process. To take the time into account that is necessary for the process of behavioural change RÜCKGEWINN is planned for duration of six months in one session weekly for 26 weeks.
  Arms: c) RÜCKGEWINN

SUMMARY:
Background:

In chronic back pain, rehabilitation specific aftercare programs, needed for a long-term improvement of pain and functional ability, are absent. Purposeful and differentiated aftercare treatments offer the possibility, in particular in the rehabilitation of chronic back pain, to increase the sustainability of positive effects of a mostly three weeks taking rehabilitation or to intensify them.

Hypothesis:

The implementation of a developed bio-psycho-social aftercare intervention program for CLBP (RÜCKGEWINN) leeds to a better rehabilitation outcome in comparison to current usual aftercare (IRENA) and a control group in view of pain-conditioned functional ability and back pain episodes.

Methods/Design:

A multicenter prospective 3-armed randomised controlled trial is conducted. 456 participants will be consecutively enrolled in inpatient and outpatient rehabilitation and assigned to either one of the three study arms. Outcomes are measured before and after rehabilitation and twelve month after dismissal form rehabilitation into the aftercare program.

DETAILED DESCRIPTION:
Background:

There is strong internationally confirmed evidence for short-term effectiveness of multimodal interdisciplinary specific treatment programmes for chronic back pain. Indeed, the proof of a lasting protection of achieved effects is missing so far. For a long-term improvement of pain and functional ability high intervention intensity or high extent seems to be necessary (> 100 therapy hours). Especially in chronic back pain rehabilitation specific aftercare programs are absent. Purposeful and differentiated aftercare treatments offer the possibility, in particular in the rehabilitation of chronic back pain, to increase the sustainability of positive effects of a mostly three weeks taking rehabilitation or to intensify them.

Hypothesis:

The implementation of a bio-psycho-social exercise based aftercare intervention program, specifically structured for the needs of chronic low back pain (CLBP) patients, leeds to a better rehabilitation outcome in comparison to current usual aftercare (IRENA) and a control group that is given an educational booklet in view of pain-conditioned functional ability and back pain episodes.

Methods/Design:

A multicenter prospective 3-armed randomised controlled trial is conducted. 456 participants will be consecutively enrolled in inpatient and outpatient rehabilitation and assigned to either one of the three study arms. Outcomes are measured before and after rehabilitation and twelve month after dismissal form rehabilitation into the aftercare program.

Discussion:

Special methodological and logistic challenges are to be mastered in this trial, which accrue from the engagement of aftercare interventions to their residential district and the fact the fact that the proportion of patients, who take part in aftercare programs, is low. The usability of the aftercare program lies in the transference into the routine care and is also given by developed manuals with structured contents, media and material for organisation assistance as well as training draughts for practise therapists in the aftercare.

ELIGIBILITY:
Inclusion Criteria:

ICD-10 is used:

* M51.2 - M51.4
* M51.8 - M51.9
* M53.8 - M53.9
* M54.5, M54.8 - M54.9
* M54.4 (if radicular symptoms are not dominating)

Exclusion Criteria:

* specific reason for back pain, based on a clear cause or diagnosis, which could sufficiently explain its extent (e.g. radicular symptomatic, myelopathesis, inflammatory changes in the spinal column etc.)
* already carried out operation on the spine within the last year
* additional serious psychic diagnosis
* uncorrected serious visual and acoustic disability
* seriously reduced health status (other diseases) with considerable reduction of dexterity
* application for retirement
* low German language skills (to fulfill the questionnaires)
* age lower than 18 or over 65
* residential area out of Berlin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Perceived pain-related functional disability as measured with the Hanover Functional Ability Questionnaire (Kohlmann & Raspe, Rehabilitation. 1996;35:I-VIII.) | one year

SECONDARY OUTCOMES:
Graded chronic pain (GCPS, Von Korff et al. 1992) | one year
Catastrophizing (KPI-AE KRSS, Hasenbring 1994) | one year
Fear avoidance Beliefs (TSK-DE, Schaub et al. 2004) | one year
Physical activity (Freiburger FB, Frey et al. 1999) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pfeifer, Prof. Dr., Principal Investigator — Institute of Sport Science and Sport / University of Erlangen-Nürnberg; Christian Hentschke, Dipl. Sportwiss., Study Director — Institute of Sport Science and Sport / University of Erlangen-Nürnberg
Locations (6):
- Germany (6):
  - Rehabilitationsklinik Lautergrund, Bad Staffelstein, Bavaria
  - Rehabilitationsklinik Dübener Heide, Bad Schmiedeberg, Brandenburg
  - MEDIAN Klinik Hoppegarten, Hoppegarten (Mark), Brandenburg
  - Zentrum für ambulante Rehabilitation (ZaR) Abt. I BO, Berlin, State of Berlin
  - Vivantes Rehabilitation Abt. I BO, Berlin, State of Berlin
  - REHA-Tagesklinik im Forum Pankow, Berlin, State of Berlin

REFERENCES:
- [Derived] Hentschke C, Hofmann J, Pfeifer K. A bio-psycho-social exercise program (RUCKGEWINN) for chronic low back pain in rehabilitation aftercare--study protocol for a randomised controlled trial. BMC Musculoskelet Disord. 2010 Nov 17;11:266. doi: 10.1186/1471-2474-11-266. PMID 21083918